CLINICAL TRIAL: NCT01814397
Title: Prospective Pilot Study to Determine the Effect of Aromatase Inhibitor-induced Estrogen Depletion on Evoked Pain Threshold and Psychosocial Factors in Breast Cancer Patients
Brief Title: Pilot Study to Evaluate the Effect of Aromatase Inhibitor Therapy on Pain Threshold in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Damon Runyon Cancer Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2008.101; HUM00026034 (Other: University of Michigan Comprehensive Cancer Center)
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Pain; Arthralgia
Keywords: Aromatase inhibitor; Pain threshold
MeSH Terms: conditions — Breast Neoplasms; Pain; Arthralgia | interventions — Anastrozole; exemestane; Letrozole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Baseline: whole blood for DNA, serum, plasma 3 month: serum, plasma 6 month: serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Women starting AI therapy: There is only a single cohort. Postmenopausal women with ER positive breast cancer who are starting treatment with anastrozole 1 mg daily, letrozole 2.5 mg daily, or exemestane 25 mg daily. Choice of therapy is at the discretion of the treating physician.
  Interventions: Drug: Anastrozole; Drug: exemestane; Drug: letrozole

INTERVENTIONS:
Drug: Anastrozole — 1 mg orally daily
  Other Names: Arimidex
Drug: exemestane — 25 mg orally daily
  Other Names: Aromasin
Drug: letrozole — 2.5 mg orally daily
  Other Names: Femara

SUMMARY:
Postmenopausal women who have hormone receptor positive breast cancer are typically treated with aromatase inhibitor medications, which substantially decrease the amount of estrogen produced by their bodies. These medications are fairly well tolerated, but can cause aches and pains which can be quite severe in some cases.

People experience pain differently. Estrogen appears to play a role in how we experience pain. Therefore, decreasing estrogen levels may lead to more pain in some women than others. The goal of this study is to evaluate perception of pain in women with breast cancer, and to determine if differences in pain perception lead to more aches and pains in some women treated with aromatase inhibitors.

In this study, we plan to enroll 55 women with breast cancer who are starting treatment with an aromatase inhibitor. Participants will undergo testing to evaluate their perception of pain, and will also complete a set of questionnaires. Testing will be conducted before starting aromatase inhibitor therapy, as well as after 3 and 6 months of therapy. We will investigate whether pre-existing differences in pain perception lead to different amounts of pain during aromatase inhibitor therapy.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Postmenopausal, age 21 or greater
* Stage 0-III estrogen receptor and/or progesterone receptor positive breast cancer who will be receiving a standard dose of letrozole, anastrozole, or exemestane
* Performance status 0-2
* Willing to sign the consent form

Exclusion Criteria:

* Average pain >=8/10 over the past 24 hours
* Peripheral sensory neuropathy grade 2 or higher
* Personal history of schizophrenia, or suicidal ideation or attempt within the past 2 years
* Thumbnail abnormalities on either hand that are likely to alter pain perception during testing

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with ER positive early stage breast cancer who are starting AI therapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norah L Henry, MD, PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Henry NL, Conlon A, Kidwell KM, Griffith K, Smerage JB, Schott AF, Hayes DF, Williams DA, Clauw DJ, Harte SE. Effect of estrogen depletion on pain sensitivity in aromatase inhibitor-treated women with early-stage breast cancer. J Pain. 2014 May;15(5):468-75. doi: 10.1016/j.jpain.2014.01.487. Epub 2014 Jan 22. PMID 24462504

RESULTS

PARTICIPANT FLOW:
Groups:
- Women Starting AI Therapy: There is only a single cohort. Postmenopausal women with hormone receptor positive breast cancer who are starting treatment with anastrozole 1 mg daily, letrozole 2.5 mg daily, or exemestane 25 mg daily. Choice of therapy is at the discretion of the treating physician.
Period: Overall Study
Arm/Group | Women Starting AI Therapy
Started | 50
3 Month Evaluation | 43
Completed | 36
Not Completed | 14
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Groups:
- Women Starting Aromatase Inhibitor (AI) Therapy: There is only a single cohort. Postmenopausal women with estrogen receptor positive breast cancer who are starting treatment with anastrozole 1 mg daily, letrozole 2.5 mg daily, or exemestane 25 mg daily. Choice of therapy is at the discretion of the treating physician.
Arm/Group | Women Starting Aromatase Inhibitor (AI) Therapy
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 60 [38 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 47
  More than one race | 0
  Unknown or Not Reported | 0
Weight, kg [Mean (Standard Deviation); unit: kilograms] | 80.7 (17.8)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 30.0 (6.5)
Aromatase inhibitor [Number; unit: participants]
  anastrozole 1 mg daily | 40
  exemestane 25 mg daily | 1
  letrozole 2.5 mg daily | 9
Prior chemotherapy [Number; unit: participants]
  prior chemotherapy | 23
  no prior chemotherapy | 27
Prior tamoxifen [Number; unit: participants]
  prior tamoxifen | 14
  no prior tamoxifen | 36
Mean Pain50, kg/cm^2 [Mean (Standard Deviation); unit: kg/cm^2] — Patients rated the intensity of each pressure sensation using a 0 to 100 numerical rating scale (0 = no pain, 100 = worst pain imaginable). Pain50 was defined as the amount of applied pressure in kilograms per square centimeter that evoked a pain intensity rating of 50 out of 100.
  kg/cm^2 | 4.3 (1.5)
Mean conditioned pain modulation (CPM) [Mean (Standard Deviation); unit: units on a scale (0-100 pain scale)] — Pressure equivalent to the patient's Pain50 was applied to the non-dominant thumbnail for 30 seconds (test stimulus), and the patient rated the intensity of the pressure on a 0-100 pain scale at 10 second intervals. Ten minutes later pressure (conditioning stimulus) was continuously applied to the dominant thumbnail for 60 seconds at the same Pain50 intensity. After 30 seconds, the test stimulus was again applied to the non-dominant thumbnail for 30 seconds and the patient rated the intensity every 10 seconds. CPM magnitude was calculated as the difference of the means of the 3 pain ratings.
  units on a scale (0-100 pain scale) | 7.9 (14.7)
Mean serum estradiol, pg/ml [Mean (Standard Deviation); unit: pg/ml] | 6.0 (7.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain50 Assessed at Baseline, 3 Months and 6 Months
Description: Patients rated the intensity of each pressure sensation using a 0 to 100 numerical rating scale (0 = no pain, 100 = worst pain imaginable). Pain50 was defined as the amount of applied pressure in kilograms per square centimeter that evoked a pain intensity rating of 50 out of 100. Pain50 was assessed at baseline, 3 months, and 6 months. Change in Pain50 with estrogen depletion was determined.
Time Frame: Baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: kg/cm^2
Arm/Group | Women Starting AI Therapy
Number analyzed (Participants) | 50
kg/cm^2
  Baseline | 4.3 (1.5)
  3 month | 4.2 (1.8)
  6 month | 4.2 (1.6)

2. Secondary Outcome: Mean Conditioned Pain Modulation Assessed at Baseline, 3 Months, and 6 Months
Description: To assess conditioned pain modulation, pressure equivalent to the patient's Pain50 was applied to the non-dominant thumbnail for 30 seconds (test stimulus), and the patient rated the intensity of the pressure on a 0-100 pain scale at 10 second intervals. Ten minutes later pressure (conditioning stimulus) was continuously applied to the dominant thumbnail for 60 seconds at the same Pain50 intensity. After 30 seconds, the test stimulus was again applied to the non-dominant thumbnail for 30 seconds and the patient rated the intensity every 10 seconds. Conditioned pain modulation magnitude was calculated as the difference (second minus first) in the mean of the 3 pain ratings to the test stimulus applied prior to and during the conditioning stimulus. Conditioned pain modulation was assessed at baseline, 3 months, and 6 months. Change over that time period was assessed. Higher conditioned pain modulation values indicate less efficient conditioned pain modulation.
Time Frame: Baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale (0-100 pain scale)
Arm/Group | Women Starting AI Therapy
Number analyzed (Participants) | 50
units on a scale (0-100 pain scale)
  baseline | 7.9 (14.7)
  3 months | 6.3 (18.4)
  6 months | 10.4 (18.9)

3. Other Pre Specified Outcome: Mean Baseline Patient-reported Symptom Measures for Patients Who Were Persistent and Nonpersistent With Aromatase Inhibitor Therapy During the First 6 Months of Treatment
Description: Patients completed 4 measures at baseline, before aromatase inhibitor therapy initiation. (1) Depression: Center for Epidemiologic Studies-Depression, scores 0-60, higher scores reflect more depression. (2) Pain: 7 day Pain Diary, scores 0-10, higher scores reflect more pain. (3) Fatigue: Multidimensional Fatigue Inventory, scores 4-20, higher scores reflect more fatigue. (4) Sleep: Medical Outcomes Study-Sleep, scores 0-100, higher scores reflect worse sleep. Persistence with aromatase inhibitor therapy was assessed at the 6 month timepoint. Mean baseline values for each measure were calculated for the cohort that persisted with aromatase inhibitor therapy and the cohort that was non-persistent.
Time Frame: Baseline patient-reported outcomes measures, 6 month persistence with therapy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Women Starting AI Therapy
Number analyzed (Participants) | 50
units on a scale
  Baseline depression, discontinuation by 6 mo | 14 (9.5)
  Baseline depression, no discontinuation by 6 mo | 6.6 (5.9)
  Baseline sleep, discontinuation by 6 mo | 47.1 (17.9)
  Baseline sleep, no discontinuation by 6 mo | 28.6 (17.8)
  BL general fatigue, discontinuation by 6 mo | 16.9 (3.6)
  BL general fatigue, no discontinuation by 6 mo | 10.6 (4.1)
  BL pain, discontinuation by 6 mo | 1.9 (1.2)
  Baseline pain, no discontinuation by 6 mo | 1.6 (1.3)

4. Other Pre Specified Outcome: Estradiol Concentration Assessments at Baseline and After 3 Months of Aromatase Inhibitor Therapy
Description: Estradiol is being assessed using an ultrasensitive gas chromatography tandem mass spectroscopy-based assay. The lower limit of detection of the assay is 0.625 pg/ml. For patients whose serum estradiol concentrations were below the lower limit of detection, the value of 0.625 pg/ml was used to calculate the mean estradiol concentration and standard deviation at both baseline and 3 months.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Women Starting AI Therapy
Number analyzed (Participants) | 50
pg/ml
  Baseline | 6.0 (7.6)
  3 months | 0.75 (0.45)

ADVERSE EVENTS:
Time Frame: 6 months
Description: We only collected data related to the study specific procedures, not the standard of care aromatase inhibitor medication.
Arm/Group | Women Starting AI Therapy
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No